CLINICAL TRIAL: NCT02505204
Title: Paravertebral Block With Versus Without Clonidine for Patients Undergoing Ventral Hernia Repair: A Prospective Double-blinded Randomized Study
Brief Title: PVB With vs. Without Clonidine for Ventral Hernia Repair
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 07/09/2015
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Ventral Hernia Repair
Keywords: clonidine; paravertebral block; hemodynamic stability
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Clonidine (Experimental): Will receive bilateral PVB with clonidine.
  Interventions: Other: Clonidine
- Placebo (Placebo Comparator): Will receive bilateral PVB with placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Clonidine — The anesthetic mixture will contain: lidocaine 2% 7 mL, lidocaine 2% 6 mL with epinephrine 5µg.mL-1, bupivacaine 0.5% 5 mL, and clonidine 2 mL.
  Arms: Clonidine
Other: Placebo — the same anesthetic mixture will be administrated however the clonidine will be substituted with 2 mL saline.
  Arms: Placebo

SUMMARY:
Paravertebral block (PVB) combined with light intravenous sedation was associated with a short hospital stay, less post-operative nausea and vomiting and reduced analgesic consumption compared to general anesthesia for ventral hernia repair. Given the effectiveness of PVB in the ventral hernia repair, it would be beneficial to study the effect of PVB with versus without clonidine in elderly patients.

Patients will be randomly allocated to one of 2 groups with 30 patients in each, using the sealed envelope technique. Group one will receive PVB with clonidine while group 2 will receive PVB with placebo.

DETAILED DESCRIPTION:
Introduction

Paravertebral block (PVB) showed to be successful in both children and adults. It has been reported to be an excellent pain reliever and it reduces post-operative nausea and vomiting, in patients undergoing breast surgery. PVB has proven to be very useful as a regional anesthetic technique when it comes to surgeries involving lumbar and thoracic dermatome. It was shown that the PVB combined with light intravenous sedation was associated with a short hospital stay, less post-operative nausea and vomiting (PONV) and reduced analgesic consumption compared to general anesthesia for ventral hernia repair. Given the effectiveness of PVB in the ventral hernia repair, it would be beneficial to study the effect of PVB with versus without clonidine in elderly patients.

Objectives:

The primary objective of this study is to compare the hemodynamic stability in a ventral hernia repair using paravertebral block with clonidine versus the PVB without clonidine.

The secondary objectives include a comparison of PONV and postoperative analgesic consumption.

Materials and Methods

Study design and sampling This is a prospective study with a randomized double- blinded design that will be conducted between August 2015 and August 2016.

Patients scheduled for ventral hernia repair whose age is 65 years and older with American Society of Anesthesiologists (ASA) greater or equal to 2 will be included. Exclusion criteria comprised history of allergic reactions to local anesthetics, bleeding diatheses and spinal abnormality.

Patients will be randomly allocated to one of 2 groups with 30 patients in each, using the sealed envelope technique. Group one will receive PVB with clonidine while group 2 will receive PVB with placebo.

Anesthetic techniques Since this trial is double-blinded, a specialized nurse will prepare the syringes for each patient.

Paravertebral nerve block techniques Bilateral nerve-stimulator PVB will be performed at the levels of T9-T10 or T9-T11 according to the type of ventral hernia and the planned incision type. The patient will be anesthetized in the lateral decubitus position. Supplemental oxygen will be given by facemask and regular anesthetic monitors will be attached.

Each local anesthetic mixture will contain:

For group 1, the syringes will contain: lidocaine 2% 6 mL, lidocaine 2% 6 mL with epinephrine 5µg.mL-1, bupivacaine 0.5% 5 mL, fentanyl 1 mL (50µg) and clonidine 2 mL.

As for the group 2, the same anesthetic mixture will be administrated however the clonidine will be substituted with 2 mL saline.

Data collection

Demographic data, ASA score, type and duration of surgery will be recorded. Haemodynamics will be registered such as the mean arterial blood pressure, heart rate and oxygen saturation, preoperatively (baseline), intra-operatively (incision of skin, dissection of hernia, traction over the sac and closure of incision) and postoperatively.

As for postoperative analgesia consumption, patients with a VAS score between three and four are given Tramadol Hydrochloride 50-100 mg every 4- 6 hours. If the VAS score is greater or equal to five, patients receive 1 mg/kg Dolosal.

Post-operative nausea and vomiting will be recorded in the recovery room and in the regular ward. Pain assessment will be taken from patients by a verbal statement using Numeric Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ventral hernia repair whose age is 65 years and older
* and with ASA greater or equal to 2

Exclusion Criteria:

* History of allergic reactions to local anesthetics
* Bleeding diatheses
* Spinal abnormality

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic stability recorded from electrocardiogram and pulse oximeter | within the first 48 hours after surgery
  Compare the hemodynamic stability between the two groups

SECONDARY OUTCOMES:
Postoperative nausea and vomiting recorded via questionnaire | within the first 48 hours after surgery
  Comparison of postoperative nausea and vomiting between the two groups
Postoperative analgesic consumption recorded via questionnaire | within the first 48 hours after surgery
  Comparison of analgesic consumption between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Chairperson of Anesthesia department
Locations (1):
- Makassed General Hospital, Beirut, Lebanon